CLINICAL TRIAL: NCT01112982
Title: Shifting the Paradigm of Gout: An Assessment of Chronic Synovial-Based Inflammation and Its Role With Serum Urate Levels.
Brief Title: An Assessment of Chronic Synovial-Based Inflammation and Its Role With Serum Urate Levels.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00000136
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2017-03

CONDITIONS: Gout
Keywords: Gout; Synovial pannus; Magnetic resonance imaging
MeSH Terms: conditions — Gout | interventions — Magnetic Resonance Spectroscopy; Febuxostat; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Febuxostat Sub-Study (Other): To analyze the effect of urate-lowering therapy (specifically with febuxostat [Uloric]) on the synovial pannus in the "index joint" of a subgroup of patients. Subjects not currently on any urate-lowering therapy, or on a serum urate lowering drug other than febuxostat (Uloric) and who have a serum urate level of > or = to 9.0, will be treated with febuxostat (Uloric) and their serum urate level will be followed at months 1, 3, 6, and 9. Magnetic Resonance Imaging (with and without gadolinium) of the same "index joint" will be repeated at month 9 to assess for the presence and degree of synovial pannus. Because initiation of urate-lowering therapy can induce acute attacks of gout, these subjects will also be started on colchicine as a prophylactic (and remain on colchicine for 6 months).
  Interventions: Other: Magnetic Resonance Imaging; Drug: Febuxostat; Drug: Colchicine
- MRI of index joint (Other): To analyze synovial pannus in the Magnetic Resonance Imaging (with and without gadolinium) of the "index joint" on Subjects not currently on any urate-lowering therapy, or on a serum urate lowering drug other than febuxostat (Uloric).
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — An Magnetic Resonance Imaging (with and without gadolinium contrast) of index joint will be performed (T1, T2, and STIR images).
  Other Names: 3 Tesla Magnetic Resonance Imaging
Drug: Febuxostat — All subjects in the sub-study will be started on febuxostat 40mg daily at baseline. If their serum urate level is > 6.0 at months 1 or 3, then the febuxostat dose will be increased to 80mg daily.
  Other Names: Uloric
  Arms: Febuxostat Sub-Study
Drug: Colchicine — Colchicine will be dosed at 0.6mg by mouth BID for the first three months then 0.6mg daily from months 3 to 6, and then discontinued at month 6.
  Other Names: Colcrys
  Arms: Febuxostat Sub-Study

SUMMARY:
The purpose of this study is to show that patients with gout suffer from chronic inflammation of their joints, observable by MRI, even in the absence of symptomatic gouty attacks. Secondary end-points of this study will include analyzing the effects of uric acid-lowering therapy (specifically with the FDA approved medication Febuxostat) in a subgroup of patients, checking for the presence of inflammatory markers to see if there is any correlation with the proposed chronic inflammation, and evaluating for other characteristic findings of gout on MRI.

DETAILED DESCRIPTION:
The clinical history of untreated gout transitions from an acute intermittent arthritis to a chronic inflammatory arthritis. This tells us that at some point the inflammation associated with gout does not abate. Our group recently completed an advanced imaging study in patients with early gout that suggested nearly 60% of subjects had synovial pannus during intercritical gout. This is likely more prevalent in patients with more advanced gout. The presence of synovial pannus also likely correlates with serum urate levels. The primary aim of this study will be to determine the percentage of patients with known gout who have evidence of chronic ongoing synovial-based inflammatory disease, determine the degree of this inflammation, and correlate it with their serum urate levels. Secondary endpoints will include assessments for the presence of other characteristic findings of gout on these MRI (i.e. erosive changes, intraosseous tophi, soft tissue tophi, joint effusion, bone marrow edema, and soft tissue edema). We will also be checking serum high-sensitivity CRP levels to evaluate for any correlation with synovial pannus, and assess baseline radiographs of the "index" joint for the presence of erosive changes, which will be correlated with the presence and severity of synovial pannus in that same joint. Analysis will also be performed to see if there is a correlation with serum urate levels. A sub-study will be performed assessing the effect of aggressive serum urate lowering therapy (specifically with febuxostat [Uloric]) on this chronic inflammation; i.e. synovial pannus.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 - Open ended to both males and females.
2. Have a known history of gout diagnosed by current or previous documentation of intracellular MSU crystals in synovial fluid, a tophus proved to contain MSU crystals, or at least six of the twelve ACR diagnostic criteria for gout (see appendix with the 12 diagnostic criteria of gout).
3. English of Spanish speaking
4. Able to give informed consent

Exclusion Criteria:

1. Age < 18.
2. Unable to give informed consent.
3. Do not speak or write in English or Spanish.
4. History of any other inflammatory arthritis.
5. History of another crystal induced arthritis.
6. Serum creatinine >1.8 mg/dL
7. Patients taking oral corticosteroids (any dose) [or within 4 weeks]
8. Parenteral or intraarticular corticosteroids within 6 weeks
9. Allergy to gadolinium contrast dye
10. Any contraindication to receiving a MRI
11. Pregnant women
12. Allergy to febuxostat (Uloric) or colchicine [substudy subjects only]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto J Rodriguez, MD, Study Director — University Of South Florida, Department of Rheumatology; John D Carter, MD, Principal Investigator — University Of South Florida, Department of Rheumatology
Locations (1):
- University of South Florida Medical Clinics, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medline Plus: Gout — http://www.nlm.nih.gov/medlineplus/ency/article/000422.htm
- See also: Medline Plus: Febuxostat — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a609020.html
- See also: Medline Plus: Colchicine — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a682711.html
- See also: Medline Plus: MRI — http://www.nlm.nih.gov/medlineplus/mriscans.html

RESULTS

PARTICIPANT FLOW:
Groups:
- MRI of Index Joint: All study participants: Standard demographics will be obtained including a baseline serum urate, creatinine, and hs-CRP. Study subjects will have their "index joint" determined (the joint that is most often involved with acute attacks of gout in each particular patient). A plain radiograph of the "index joint" will be obtained, as well as an MRI with and without gadolinium enhancement to assess for presence and degree synovial pannus.
  Magnetic Resonance Imaging: An MRI (with and without gadolinium contrast) of index joint will be performed (T1, T2, and STIR images).
  Plain Radiographs: Plain radiographs of "index joint" will be obtained and reviewed by two independent readers (radiologists)
Period: Overall Study
Arm/Group | MRI of Index Joint
Started | 74
Completed | 72
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — exceeded weight limit to complete MRI | 1

BASELINE CHARACTERISTICS:
Arm/Group | MRI of Index Joint
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 67
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 56.4 [28 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 59
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Evidence of Chronic Ongoing Synovial-Based Inflammatory Disease at Baseline.
Description: The primary aim of this study will be to determine the percentage of patients with known gout who have evidence of chronic ongoing synovial-based inflammatory disease, i.e. synovial pannus, in their "index joint", and determine if there is a correlation of the prevalence and severity of synovial pannus in the "index joint" with the patients' serum urate levels on the day of their MRI.
Time Frame: MRI and baseline uric acid level will be performed upon enrollment in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | MRI of Index Joint
Number analyzed (Participants) | 72
Participants | 63
Statistical Analysis 1: Comparison: MRI of Index Joint; Presence of synovial pannus and the serum urate level; Test type: Other; p = 0.34, t-test, 2 sided

2. Secondary Outcome: Number and Percentage of Substudy Participants for Whom the Severity of Synovial Pannus Was Significantly Reduced After 9 Months of Treatment With Febuxostat (Uloric).
Description: A sub-study in a subgroup of patients will analyze the Number and Percentage of Substudy Participants for whom the Severity of Synovial Pannus was Significantly Reduced After 9 Months of Treatment with Febuxostat (Uloric) in the "index joint" by comparing the baseline MRI with a repeat MRI of the same joint.
Time Frame: Upon enrollment into study, and at month 9.
Measure: Count of Participants; unit: Participants
Groups:
- Febuxostat Sub-Study: The primary endpoint of this sub-study was to determine if a nine month course of aggressive serum ULT in patients with gout significantly affects the severity of synovial pannus in the index joint as determined by comparing the baseline and month 9 MRI's using the aforementioned grading scale. Secondary endpoints included an assessment of significant change of the subjects' serum CRP and estimated Glomerular Filtration Rate (eGFR) from baseline to month 9. Other endpoints included assessing for significant change of erosive changes, intraosseous tophi, soft tissue tophi, joint effusion, bone marrow edema/lesions, and soft tissue edema on the MRI from baseline to month 9.
Arm/Group | Febuxostat Sub-Study
Number analyzed (Participants) | 32
Participants | 25

3. Secondary Outcome: Number of Participants With Other Characteristic Findings of Gout on MRI's Correlated With Serum Urate Levels.
Description: Number of Participants with Other Characteristic Findings of Gout on these MRI's. These include erosive changes, intraosseous tophi, soft tissue tophi, joint effusion, bone marrow edema, and soft tissue edema. These secondary endpoints will also be summed with patients' serum urate levels.
Time Frame: Upon enrollment into study
Measure: Count of Participants; unit: Participants
Arm/Group | MRI of Index Joint
Number analyzed (Participants) | 72
Participants
  Erosive Changes | 31
  Intraosseous tophi | 25
  Soft tissue tophi | 11
  Joint effusion | 14
  Bone marrow edema | 40
  Soft tissue edema | 28
Statistical Analysis 1: Comparison: MRI of Index Joint; The Severity of Synovial Pannus and the Serum Urate level; Test type: Other — Spearman Correlation Coefficient; p = 0.73, t-test, 1 sided

4. Secondary Outcome: Mean Serum Urate Levels for Previous 2 Years at Baseline.
Description: Determine if there is a correlation between the prevalence and severity of synovial pannus in the "index joint" with the patients' mean serum urate level from the previous 2 years at baseline.
Time Frame: previous 2 years upon enrollment into study
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- MRI of Index Joint: To analyze synovial pannus in the Magnetic Resonance Imaging (with and without gadolinium) of the "index joint" on Subjects not currently on any urate-lowering therapy, or on a serum urate lowering drug.
  Magnetic Resonance Imaging: An Magnetic Resonance Imaging (with and without gadolinium contrast) of index joint will be performed (T1, T2, and STIR images).
Arm/Group | MRI of Index Joint
Number analyzed (Participants) | 72
mg/dL | 7.93 (2.13)
Statistical Analysis 1: Comparison: MRI of Index Joint; Test type: Other — correlation between severity of synovial pannus and the serum urate level; p = 0.73, t-test, 1 sided

5. Secondary Outcome: The Severity of Synovial Pannus the Day of Serum High-sensitivity C-Reactive Protein and Magnetic Resonance Imaging
Description: Determine if the Number of Participants Prevalence and Severity of Synovial Pannus in the "Index Joint" with the patient's serum high-sensitivity C-Reactive Protein on the same day as the Magnetic Resonance Imaging. The Magnetic Resonance Imaging will be assessed for the severity of synovial pannus, which is graded on a scale of 1 to 6 (with 6 being the most severe).
Time Frame: Upon enrollment into study at screening.
Population: Severity of Synovial Pannus in the "Index Joint"
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MRI of Index Joint | Febuxostat Sub-Study
Number analyzed (Participants) | 72 | 25
units on a scale | 2.99 (1.3) | 3.42 (1.3)
Statistical Analysis 1: Comparison: MRI of Index Joint; Test type: Other; p = 0.32, t-test, 1 sided — The presence of synovial pannus in the "index joint"

6. Secondary Outcome: Presence or Absence of Erosive Changes on Baseline Radiographs of the "Index" Joint Correlated With the Presence and Severity of Synovial Pannus Correlation With Serum Urate Levels and the Presence of Erosions on Their Plain Radiograph.
Description: Baseline radiographs of the "index" joint will also be obtained on the same day as their MRI and assessed for the presence or absence of erosive changes, intraosseous tophi, soft tissue tophi, joint effusion, bone marrow edema, or soft tissue edema. This will be correlated with the presence and severity of synovial pannus in that same joint. The analysis will also be performed to see if there is a correlation with serum urate levels and the presence of erosions on their plain radiograph.
Time Frame: Upon enrollment into study
Measure: Count of Participants; unit: Participants
Arm/Group | MRI of Index Joint
Number analyzed (Participants) | 72
Participants
  Erosive Changes: Presence | 31
  Erosive Changes: Absence | 41
  Serum urate levels ≤6.8mg/dL: Presence | 24
  Serum urate levels ≤6.8mg/dL: Absence | 48
  Intraosseous Tophi: Presence | 25
  Intraosseous Tophi: Absence | 47
  Soft Tissue Tophi: Presence | 11
  Soft Tissue Tophi: Absence | 61
  Joint Effusion: Presence | 14
  Joint Effusion: Absence | 58
  Bone Marrow Edema: Presence | 40
  Bone Marrow Edema: Absence | 32
  Soft Tissue Edema: Presence | 28
  Soft Tissue Edema: Absence | 44
Statistical Analysis 1: Comparison: MRI of Index Joint; The absence of erosive changes; Test type: Other — Kappa Coefficient; p = 0.09, t-test, 2 sided
Statistical Analysis 2: Comparison: MRI of Index Joint; Test type: Other — the absence of Intraosseous Tophi; p = 0.33, t-test, 2 sided
Statistical Analysis 3: Comparison: MRI of Index Joint; Test type: Other — The absence of Soft Tissue Tophi; p = 0.09, t-test, 2 sided
Statistical Analysis 4: Comparison: MRI of Index Joint; Test type: Other — The absence of Joint Effusion; p = 0.31, t-test, 2 sided
Statistical Analysis 5: Comparison: MRI of Index Joint; Test type: Other — The absence of Bone Marrow Edema; p = 0.25, t-test, 2 sided
Statistical Analysis 6: Comparison: MRI of Index Joint; Test type: Other — The absence of Soft Tissue Edema; p = 0.14, t-test, 2 sided

7. Secondary Outcome: High-sensitivity C-Reactive Protein Concentrations
Description: The concentration of serum high-sensitivity C-Reactive Protein at enrollment.
Time Frame: Upon enrollment into study at screening.
Population: Serum High-Sensitivity C-Reactive Protein
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MRI of Index Joint | Febuxostat Sub-Study
Number analyzed (Participants) | 72 | 25
mg/dL | 0.52 (0.84) | 0.37 (0.4)
Statistical Analysis 1: Comparison: MRI of Index Joint; Test type: Other; p = 0.32, t-test, 1 sided — The Presence of synovial Pannus in the "index joint"
Statistical Analysis 2: Comparison: MRI of Index Joint; Test type: Other; p = 0.99, t-test, 1 sided — The Severity of Synovial Pannus in the "index joint"

ADVERSE EVENTS:
Time Frame: At screening, baseline, week 2, month 1, month 3, month 6, and month 9 adverse events were collected on 72 study participants.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were monitored/assessed.
Arm/Group | MRI of Index Joint
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 1/72
Other Adverse Events (participants affected / at risk) | 8/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI of Index Joint (N=72)
exacerbation of congestive heart failure (Cardiac disorders) | 1 (1) — exacerbation of congestive heart failure requiring hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI of Index Joint (N=72)
increased liver function tests (Hepatobiliary disorders) | 8 (8) — increased liver function tests (LFT). 8/25 (32%) subjects experienced some degree of LFT elevation during the study, but only 1 (4%) subject experienced increased LFTs of greater than two times the upper limit of normal.
thrombocytopenia (Cardiac disorders) | 1 (1) — mild thrombocytopenia without complication.
mild nausea (Gastrointestinal disorders) | 2 (2) — experienced mild nausea that resolved with supportive care.

LIMITATIONS AND CAVEATS:
two subjects who did not complete the entire protocol, one exceeded the weight limit to complete the MRI, and the other withdrew consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No